CLINICAL TRIAL: NCT02972060
Title: A Phase 2 Randomized Open-Label Study of Oral Darolutamide (ODM-201) vs. Androgen Deprivation Therapy (ADT) With LHRH Agonists or Antagonist in Men With Hormone Naive Prostate Cancer
Brief Title: ODM-201 vs Androgen Deprivation Therapy in Hormone naïve Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1532; 2016-004334-17 (EudraCT Number)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Hormone Naive Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADT (Active Comparator): The standard treatment for this stage of the disease is ADT by means of LHRH antagonist for 24 weeks or by LHRH agonist therapy for 24 weeks with 4 weeks of anti-androgen to prevent flare.
  This includes leuprolide, goserelin, triptorelin, and degarelix. Beyond week 24, the treatment will be left to the discretion of the treating physician.
  Interventions: Drug: ADT
- ODM 201 (Experimental): ODM 201 will be administered as oral 300-mg tablets. The dose of study drug to be administered is 600 mg (2 x 300-mg tablets) bid for a daily dose of 1200 mg. It is recommended that ODM-201 be taken with food.
  Subjects who have clinical benefit at week 24 may continue to receive ODM-201 at the discretion of the investigator until disease progression, objective or clinical, or occurrence of an unacceptable toxicity. This includes those that will receive external beam radiation therapy.
  Any anti-cancer therapy other than the study drug given as single agent will not be considered part of the protocol treatment.
  Interventions: Drug: ODM-201

INTERVENTIONS:
Drug: ODM-201 — ODM-201 is a novel, oral, potent nonsteroidal AR inhibitor. ODM 201 will be administered as oral 300-mg tablets. The dose of study drug to be administered is 600 mg (2 x 300-mg tablets) b.i.d. to a daily dose of 1200 mg. It is recommended that ODM-201 be taken with food. Treatment should be initiated within 28 days from randomization.
  Arms: ODM 201
Drug: ADT — ADT by means of LHRH antagonist for 24 weeks or by LHRH agonist therapy for 24 weeks with 4 weeks of anti-androgen to prevent flare.
  This includes leuprolide, goserelin, triptorelin, and degarelix. Beyond week 24, the treatment will be left to the discretion of the treating physician.
  Arms: ADT

SUMMARY:
This is an open label non-comparative controlled randomized phase II study. The experimental arm is the group receiving ODM-201. The group receiving androgen-deprivation therapy (ADT) is included as an internal control.

The primary trial objective is to demonstrate that ODM-201 produces prostate-specific antigen (PSA) response rates at 24 weeks (defined as ≥80% reduction compared to baseline) that are in the range of those achieved with 24 weeks of ADT.

In total, this 1:1 randomized study will therefore require randomization of at least 250 patients, 125 to each arm.

DETAILED DESCRIPTION:
ODM 201 will be administered as oral 300-mg tablets. The dose of study drug to be administered is 600 milligrams (mg) (2 x 300-mg tablets) twice daily (bid) for a daily dose of 1200 mg. It is recommended that ODM-201 be taken with food.

Subjects who have clinical benefit at week 24 may continue to receive ODM-201 at the discretion of the investigator until disease progression, objective or clinical, or occurrence of an unacceptable toxicity. This includes those that will receive external beam radiation therapy.

Any anti-cancer therapy other than the study drug given as single agent will not be considered part of the protocol treatment.

The standard treatment for this stage of the disease is androgen deprivation therapy (ADT) by means of Luteinizing hormone-releasing hormone (LHRH) antagonist for 24 weeks or by LHRH agonist therapy for 24 weeks with 4 weeks of anti-androgen to prevent flare.

This includes leuprolide, goserelin, triptorelin, and degarelix. Beyond week 24, the treatment will be left to the discretion of the treating physician.

The primary trial objective is to demonstrate that ODM-201 produces prostate-specific antigen (PSA) response rates at 24 weeks (defined as ≥80% reduction compared to baseline) that are in the range of those achieved with 24 weeks of ADT.

The secondary objectives are to:

* To document the effects of ODM-201 compared to ADT in terms of patient-reported side effects of hormonal therapy, based on the Hormonal treatment (HTR) symptom scale of EORTC QLQ PR25 at 24 weeks;
* To document the effects of ODM-201 compared to ADT in terms of patient-reported side effects of hormonal therapy, based on EORTC QLQ C30 and PR25 at 24 weeks;
* To document the effect of ODM-201 on PSA complete response at 24 weeks (defined as ≥ 90% reduction from baseline);
* To document the effect of ODM-201 on objective response rate at 24 weeks in patients with RECIST 1.1 measurable disease at baseline;
* To document the safety and tolerability of ODM-201 vs. ADT in subjects who have not previously received hormone treatment for prostate cancer;
* To document the effects of ODM-201 on androgen deprivations symptoms using the Aging male symptoms (AMS) questionnaires;
* To document the proportion of patients who opted to continue treatment with ODM-201 beyond the protocolized 24 weeks

The primary endpoint is the PSA response assessed at 24 weeks. PSA response is defined as a ≥ 80% decline in PSA measurement taken at week 24 relative to the measurement taken at baseline, in the ODM-201 study arm. The ADT arm is used as an internal control.

Key secondary endpoints:

* Change in hormone-treatment related symptoms scale of the EORTC QLQ-PR25 at 24 weeks compared to baseline in the ODM-201 study arm. A 10-point difference is regarded as a clinically meaningful benefit.
* Objective response rate at 24 weeks in patients with RECIST 1.1 measurable disease at baseline
* PSA response at 24 weeks defined as a ≥90% decline in PSA compared to baseline
* Safety according to National Cancer Institute - Common terminology for adverse events (NCI-CTC) version 4.0

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer (all stages) for whom continuous androgen-deprivation therapy (ADT) is indicated for a minimum period of 24 weeks
* Patient presenting with a maximum of 4 confirmed metastatic lesions, including bone, extra-pelvic lymph nodes, and pelvic lymph nodes > 2 cm on baseline Computed tomography(CT) or Magnetic resonance imaging (MRI) and/or Tc bone scintigraphy. Visceral metastases are excluded
* Asymptomatic for metastatic prostate cancer; urinary symptoms are allowed
* Baseline testosterone ≥ 8 nmol/L or 230 ng/dL
* Two subsequent PSA values ≥ 2 ng/ml, taken at minimum 2-week interval, with the second being equal to or higher than the first one
* WHO performance status (PS) of 0-1
* G8 score ≥ 14 for patients aged ≥ 70 years old
* A life expectancy of at least 12 months
* Able to swallow the study drug and comply with the study requirements
* Adequate bone marrow function (absolute neutrophil count (ANC) ≥ 1.5 10exp9/L; hemoglobin ≥ 10.0 g/dl, platelets ≥ 100 10exp9/L)
* Adequate renal function: creatinine clearance/eGFR within normal limits to baseline assessed as per local standard method
* Albumin > 25 g/L
* Adequate hepatic function:

Bilirubin: total bilirubin ≤ to 1.5 X upper limit of normal (ULN)

* Aspartate aminotransferase (AST) and/or Alanine aminotransferase(ALT) ≤ 2.5 X ULN
* Normal cardiac function according to local standard by 12-lead Electrocardiogram (ECG) (complete, standardized 12-lead recording)
* Before patient registration/randomization, written informed consent must be given according to International Conference on Harmonization on Good Clinical Practices (ICH/GCP), and national/local regulations.

Exclusion Criteria:

* any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Previously or currently receiving hormonal therapy with intent to treat prostate cancer disease (surgical castration or other hormonal manipulation, e.g. GnRH agonists, GnRH antagonists, anti-androgens, oestrogens, 5α-reductase inhibitor). For patients that have received (neo)adjuvant ADT before radiotherapy, it should have been stopped for more than 1 year
* Prior use of investigational agents that block androgen synthesis or block androgen receptor
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g. saw palmetto)
* Has received systemic glucocorticoids within 24 weeks prior to enrollment or is expected to require systemic glucocorticoids during the study period
* Radiation therapy for treatment of the primary tumor within 3 months prior to enrollment
* Use of an investigational agent within 4 weeks prior to enrollment is not allowed. The maximum allowed duration may be extended to comply with national regulations in the participating countries.
* Gastrointestinal disorder affecting absorption (e.g. gastrectomy, active peptic ulcer disease within 3 months prior to enrollment)
* Known hypersensitivity to the study treatment or any of its ingredients (refer to Investigator's brochure).
* Severe or uncontrolled concurrent disease, infection or co-morbidity including active viral hepatitis, known human immunodeficiency virus infection with detectable viral load (Human immunodeficiency virus (HIV)) or chronic liver disease
* History of prior malignancy. Adequately treated basal cell or squamous cell carcinoma of skin or superficial bladder cancer that has not spread behind the connective tissue layer (i.e. pTis, pTa, and pT1) is allowed, as well as any other cancer for which chemotherapy has been completed ≤ 5 years ago and from which the patient has been disease-free.
* Clinically significant cardiovascular disease including:
* Myocardial infarction within six months prior to randomization
* Uncontrolled angina within 3 months prior to randomization
* Coronary/peripheral artery bypass within 6 months prior to randomization
* Stroke within 6 months prior to randomization
* Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or subjects with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within 3 months results in a left ventricular ejection fraction that is ≥ 45%
* History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
* History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
* Uncontrolled hypertension as indicated by a resting systolic blood pressure >170 mm Hg or diastolic blood pressure > 105 mm Hg at the screening visit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
PSA response | 24 weeks
  PSA response is defined as a ≥ 80% decline in PSA measurement taken at week 24 relative to the measurement taken at baseline, in the ODM-201 study arm. The ADT arm is used as an internal control.

SECONDARY OUTCOMES:
EORTC QLQ-PR25 | 24 weeks
  Change in hormone-treatment related symptoms scale of the EORTC QLQ-PR25 at 24 weeks compared to baseline in the ODM-201 study arm. A 10-point difference is regarded as a clinically meaningful benefit.
Objective tumor response | 24 weeks
  Objective response rate at 24 weeks in patients with RECIST 1.1 measurable disease at baseline
90% PSA response rate | 24 weeks
  PSA response at 24 weeks defined as a ≥90% decline in PSA compared to baseline
evaluation of safety | The collection period will start from randomization until 30 days after last protocol treatment administration.
  All adverse events will be recorded; the investigator will assess whether those events are drug related (reasonable possibility, no reasonable possibility) and this assessment will be recorded in the database for all adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Tombal, Pr, Study Chair — Cliniques universitaires saint-Luc (Brussels)
Locations (12):
- Belgium (4):
  - Hopitaux Universitaires Bordet-Erasme - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - CHU Dinant Godinne - UCL Namur, Yvoir
- France (2):
  - CHU de Dijon - Centre Georges-Francois-Leclerc, Dijon
  - Gustave Roussy, Villejuif
- Azienda Ospedaliera Citta della Salute e della Scienza di Torino - Ospedale Molinette, Torino, Italy
- Spain (5):
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Fundacion Instituto Valenciano De Oncologia, Valencia

IPD SHARING:
Plan to Share IPD: No